CLINICAL TRIAL: NCT03073759
Title: Effect of Transcranial Direct Current Stimulation on Proprioceptive and Vibratory Sensation: Potential Benefit for Patients With Peripheral Neuropathy
Brief Title: Effect of Transcranial Direct Current Stimulation on Peripheral Neuropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00066426
Record Dates: First submitted 2016-04-01; First posted 2017-03-08 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dTCS (Experimental): Patient will receive dTCS with direct current (maximum of 2 mA) stimulation delivered through surface electrodes (TransQE from IOMED®, surface area: 25 cm2) using a Phoresor® II Auto (Model No. PM850, IOMED®, Salt Lake City, Utah 84120, USA) or Sham stimulation.
  Interventions: Device: dTCS
- Sham (Sham Comparator): Patients will receive a sham.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: dTCS — Direct current (DC) (maximum of 2 mA) stimulation delivered through surface electrodes. One electrode will be positioned above the left or right primary motor cortex, the other electrode over the forehead.
  Arms: dTCS
Device: Sham device — The device will administer a sham.
  Arms: Sham

SUMMARY:
This study will be performed in patients with peripheral neuropathy who are walking independently, but have complains of balance problems such as recent falls or difficulty walking and show reduced vibratory and proprioceptive sensation during routine neurologic examination. These patients will be tested for proprioceptive and vibratory threshold at the toes and ankles before, during and after receiving anodal direct transcranial cortical stimulation (dTCS) over sensory and motor cortices. Subjects will be asked to participate in 2 sessions.

DETAILED DESCRIPTION:
This study will be performed in patients with peripheral neuropathy who are walking independently, but have complains of balance problems such as recent falls or difficulty walking and show reduced vibratory and proprioceptive sensation during routine neurologic examination. These patients will be tested for proprioceptive and vibratory threshold at the toes and ankles before, during and after receiving anodal transcranial direct current stimulation (tDCS) over sensory and motor cortices. Subjects will be asked to participate in 2 sessions. In one of the sessions, decided randomly, the stimulation will be applied on the right side and in the second session it will be on the left.

The tDCS portion of the experiment will begins with direct current (maximum of 2 mA) stimulation delivered through surface electrodes (TransQE from IOMED®, surface area: 25 cm2) using a Phoresor® II Auto (Model No. PM850, IOMED®, Salt Lake City, Utah 84120, USA). One electrode will be positioned above the left or right primary motor cortex, the other electrode over the forehead.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Neuropathy
* Walking independently but with problems with balance

Exclusion Criteria:

* Prominent weakness at the ankle
* Not able to walk independently
* History of Seizure
* Cardiac Pacemaker
* Metal implants in the head
* Increased intracranial pressure
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Khoshnoodi, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- dTCS: patients received dTCS
- Sham: Subjects received Sham stimulation
Period: Overall Study
Arm/Group | dTCS | Sham
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dTCS | Sham | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (2) | 67 (1.6) | 65 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Vibratory Threshold as Measured by Rydel Seiffer Graduated Tuning Fork at the Toes
Description: Vibration is measured by reading in Rydel Seiffer tuning fork that ranges between 0-8 and is a standard tool fro measuring vibration sensation at the toes. A reading of 0 means absent vibration. A reading of more than 4 at the toes are considered normal. Change between assessment at 20 minutes and 10 minutes at the toes will be assessed. A recording of less than 4 indicates an abnormal results and a lower number means worse neuropathy. For example, reading of 0 means absent vibration feeling which indicates worse neuropathy than a reading of 2.
Time Frame: At 10 and 20 minutes
Population: Due to lack of participation for sham group, data for outcome measures in sham group was not collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | dTCS | Sham
Number analyzed (Participants) | 2 | 0
units on a scale | 0 (0) |

2. Primary Outcome: Change in Minimum Detectable Angle (Degree) of Dorsiflexion of the Toe
Time Frame: At 10 and 20 minutes
Population: Not enough patients were enrolled to reach the needed threshold to assess this outcome measure. Therefore, data was not collected.
Arm/Group | dTCS | Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | dTCS | Sham
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Low number of subjects prevented statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03073759/Prot_SAP_000.pdf